CLINICAL TRIAL: NCT04802291
Title: HomeStyles-2: Shaping HOME Environments and LifeSTYLES to Prevent Childhood Obesity
Acronym: HomeStyles-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Carol Byrd-Bredbenner, PhD, RD, FAND, Distinguished Professor of Nutrition, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro2020001192
Record Dates: First submitted 2021-03-14; First posted 2021-03-17 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Healthy Lifestyle; Home Environment Related Disease; Cognitive Change; Child Behavior; Child Obesity; Parenting; Parents; Parent-Child Relations
Keywords: middle childhood; parent; lifestyle; home environment; obesity; Social Cognitive Theory
MeSH Terms: conditions — Child Behavior; Pediatric Obesity; Obesity

STUDY DESIGN:
Intervention Model Description: experimental group and an attention control group
Who Masked: Participant
Masking Description: concurrent treatments different in subject matter but equal in nonspecific treatment effects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy HomeStyles (Experimental): Online educational intervention addressing salient factors affecting school-age children's health and nutritional status: inadequate intake of fruits and vegetables, infrequent family meals, excessive consumption of sugar-sweetened beverages, large portion sizes, irregular breakfast consumption, limited physical activity, and inadequate sleep as well as children's limited food preparation skills.
  Interventions: Behavioral: HomeStyles-2: Obesity Prevention Program for Families with Children in Middle Childhood
- Safe HomeStyles (Active Comparator): Online educational intervention addressing aspects of home safety issues, such as indoor air quality, mold & moisture, hazardous household products, carbon monoxide, home safety, foodborne illness, and refrigerator temperatures.
  Interventions: Behavioral: HomeStyles-2: Obesity Prevention Program for Families with Children in Middle Childhood

INTERVENTIONS:
Behavioral: HomeStyles-2: Obesity Prevention Program for Families with Children in Middle Childhood — Comparison of 2 educational interventions

SUMMARY:
Parents are children's primary role models, are food and physical activity gatekeepers, and create the structure/lifestyle environment within the home. Thus, parents strongly influence children's weight-related behaviors and have the opportunity to cultivate a "culture of health" within the home. Yet, there continues to be a dearth of evidence-based obesity prevention intervention programs, especially for families with children aged 6 to 11 years, commonly called the middle childhood years. The aim of the HomeStyles-2 online learning mode RCT is to determine whether this novel, age-appropriate, family intervention enables and motivates parents to shape their home environments and weight-related lifestyle practices (i.e., diet, exercise, sleep) to be more supportive of optimal health and reduced risk of obesity in their middle childhood youth more than those in the control condition. The RCT will include the experimental group and an attention control group who will engage in a bona fide concurrent treatment different in subject matter but equal in nonspecific treatment effects. The participants will be families with school-age children who are systematically randomly assigned by computer to study condition. The HomeStyles intervention is predicated on the social cognitive theory and a social ecological framework. The RCT will collect sociodemographic characteristics of the participant, child, and partner/spouse; child and parent health status; parent weight-related cognitions; weight-related behaviors of the parent and child; and weight-related characteristics of the home environment. Enrollment for this study will begin mid-2021.This paper describes these aspects of the HomeStyles-2 intervention: rationale; sample eligibility criteria and recruitment; study design; experimental group intervention theoretical and philosophical underpinnings, structure, content, and development process; attention control intervention; survey instrument development and components; outcome measures; and planned analyses.

DETAILED DESCRIPTION:
The aim of the HomeStyles-2 online learning mode RCT is to determine whether this novel, age-appropriate, family intervention enables and motivates parents to shape their home environments and weight-related lifestyle practices (i.e., diet, exercise, sleep) to be more supportive of optimal health and reduced risk of obesity in their middle childhood youth more than those in the control condition. RCT Design CONSORT guidelines extension for social and psychological intervention trials will be used to generate a participant flow diagram and report RCT enrollment and retention data.113 Interested participants will begin by completing a short eligibility screener survey. Eligible participants who give informed consent will have immediate access to the baseline survey. Those who complete the baseline survey, meet survey plausibility checks (e.g., consistent answers to items measuring the same concept, meet minimal likely completion time, do not answer to all questions on a survey page the same), and complete the registration page (i.e., provide name and contact information) will be enrolled in the RCT. Enrolled participants will be systematically randomized by computer by alternating assignment to the experimental or attention control study condition. Recruitment materials and the bona fide treatment to be delivered to the attention control group are designed to blind participant assignment to study condition. Participants will receive intervention materials starting immediately after registration and at weekly intervals for 8 weeks. In week 9 of the study, participants will be invited to take the post survey to assess intervention effects Approximately 8 to 10 weeks after participants complete the post survey, they will be invited to take the follow-up survey to assess longer-term intervention effects.

Each week parents will be encouraged to spend about 15 minutes reviewing intervention materials; think about the changes like those suggested in the materials that could help their families; and implement 1 or 2 easy, quick, low-cost changes in their homes. Intervention materials (described in a subsequent section) provided each week for 8 weeks include an electronic informational guide for parents, tracker to list guide-related goals for the week and monitor progress toward them, 3 to 4 encouraging nudges delivered by SMS and email, and a guide for kids that is available electronically and is mailed to the participant homes along with a reminder magnet.

Participant progress through the RCT will be monitored by project staff by observing their visits to the website. Bilingual staff will be trained in customer service strategies and instructed to quickly address any participant queries submitted by email or phone using scripted responses to ensure equitable care across study groups. Participants will receive modest stipends that increase in value after they complete each survey.

Experimental Group Intervention The HomeStyles-2 experimental group intervention materials (i.e., "Healthy" HomeStyles-2) were designed to be congruent with White House and IOM recommendations for home-centered obesity prevention interventions and critical elements for effective interventions (e.g., interventions are positive, culturally sensitive, supportive of parent-child interaction and child development; develop realistic, effective plans that empower families). Like HomeStyles for preschoolers, HomeStyles-2 for middle childhood intervention materials provide intensive, interactive, fun, non-judgmental opportunities for parents to shape their home environments and lifestyle practices to protect child health. They also promote positive strategies and changes that adults can control in their environments to reduce risk of excessive weight gain in their middle childhood youth. A positive approach teaches individuals what they can do (eat more fruits) rather than giving prohibitions (cut out fries). Substantial evidence supports parent preference for positive messages and the value of promoting positive vs restrictive behaviors to achieve health goals.

Intervention Content. Key factors contributing to childhood obesity that can be suitably addressed in the home environment with middle childhood kids identified for inclusion in the intervention materials were selected using systematic literature reviews and input from experts in childhood obesity prevention. The most salient factors affecting school-age children's health and nutritional status that emerged were inadequate intake of fruits and vegetables, infrequent family meals, excessive consumption of sugar-sweetened beverages, large portion sizes, irregular breakfast consumption, limited physical activity, and inadequate sleep. An additional factor was children's limited food preparation skills. Attitudes toward engaging in healthy behaviors (i.e., eating fruits and vegetables, having family meals, curtailing intake of sweet beverages, controlling portion sizes, eating breakfast, getting physical exercise and limiting screentime, getting sufficient sleep, and giving children food preparation opportunities), barriers to performing healthy behaviors, strategies for overcoming barriers to healthy behaviors, and confidence in the ability to perform healthy behaviors regularly, as well as determinants of quality of life, were explored via focus groups with parents of middle-childhood youth and children ages 6 to 11 years.

Attention Control Intervention The attention control intervention will use bona fide, credible materials that are structurally equivalent to the experimental group. The attention control treatment will be credible in that it focuses on a topic fitting the description of the study recruitment materials (i.e., shaping homes and lifestyles to help kids grow up even happier and healthier) yet providing distinctly different, non-overlapping content (i.e., home safety) devoid of the RCT "active" ingredient (i.e., content related to childhood obesity prevention). The attention control intervention materials include the same components as those used in the experimental group (i.e., parent guides, trackers, children's guides, and reminder magnets) with the content focused on home safety.

The Safe HomeStyles parent guides, like the HomeStyles! Guide for the experimental group provided an overview of home safety. The other parent guides, as well as the children's guides, trackers, and reminder magnets, focus on indoor air quality, mold & moisture, hazardous household products, carbon monoxide, home safety, foodborne illness, and refrigerator temperatures. The Safe HomeStyles materials have an appearance and structure similar to those in the experimental group.

Instruments The study survey, "Home Obesogenicity Measure of EnvironmentS"-Families with School-age Kids (HOMES-FSAK), will be used to collect baseline, post, and follow-up data in the HomeStyles-2 RCT. The Social Cognitive Theory along with the key concepts addressed in the HomeStyles-2 guides provided the framework for identification of cognitions, behaviors, and aspects of the home environment to be assessed. Online survey collection procedures will be used to collect baseline, post, and follow-up data. The survey will collect sociodemographic characteristics of the participant, child, and partner/spouse; child and parent health status; parent weight-related cognitions; weight-related behaviors of the parent and child; and weight-related characteristics of the home environment.

ELIGIBILITY:
Inclusion Criteria:

* parent between the ages of 24 and 50 years with at least 1 child aged 6 to 11 years; primary food gatekeeper in the household (i.e., makes all or most decisions related to family food choices), have regular Internet access, read English and/or Spanish, and reside in the United States

Exclusion Criteria:

* Does not fit inclusion criteria

Ages: 24 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 269 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Child Weight-Related behaviors | Pre-intervention (baseline), post-intervention (~8 weeks after baseline), follow-up (~4 weeks after post-intervention)
  Child dietary intake, physical activity, and sleep behaviors

SECONDARY OUTCOMES:
Parent Weight-Related Cognitions | Pre-intervention (baseline), post-intervention (~8 weeks after baseline), follow-up (~4 weeks after post-intervention)
  Parent self-efficacy, outcome expectations, attitudes, modeling
Supports for Obesity-Preventive Measures | Pre-intervention (baseline), post-intervention (~8 weeks after baseline), follow-up (~4 weeks after post-intervention)
  Parent weight-related parenting behaviors; home availability of foods; space and supports for physical activity
Parent Weight-Related behaviors | Pre-intervention (baseline), post-intervention (~8 weeks after baseline), follow-up (~4 weeks after post-intervention)
  Parent dietary intake, physical activity, and sleep behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Carol Byrd-Bredbenner, PhD, Principal Investigator — Rutgers Universitiy
Locations (1):
- Rutgers University, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Derived] Byrd-Bredbenner C, Santiago E, Eck KM, Delaney CL, Quick VM, Pozzoli A, Worobey J, Shelnutt KP, Olfert MD. HomeStyles-2: Randomized controlled trial protocol for a web-based obesity prevention program for families with children in middle childhood. Contemp Clin Trials. 2022 Jan;112:106644. doi: 10.1016/j.cct.2021.106644. Epub 2021 Dec 1. PMID 34861408